CLINICAL TRIAL: NCT03585036
Title: Oral Tramadol Versus Oral Dexketoprofen for Reducing Pain During Office Hysteroscopy in Post Menopausal Women
Brief Title: Oral Tramadol Versus Oral Dexketoprofen for Reducing Pain During Office Hysteroscopy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, lecturer in obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: tramadol
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Hysteroscopy
MeSH Terms: interventions — dexketoprofen trometamol; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- dexketoprofen (Active Comparator): Drug: dexketoprofen Women will receive oral dexketoprofen 25mg 2 hours before the procedure
  Drug: Placebo 1 Women will receive an oral placebo similar to Tramadol 2 hours before the procedure.
  Interventions: Drug: dexketoprofen
- tramadol (Active Comparator): Drug: Tramadol Women will receive oral Tramadol 100 mg 2 hours before the procedure
  Drug: Placebo 2 Women will receive an oral placebo similar to dexketoprofen 2 hours before the procedure
  .
  Interventions: Drug: Tramadol
- placebo (Placebo Comparator): Drug: Placebo 1 Women will receive an oral placebo similar to Tramadol 2 hours before the procedure.
  Drug: Placebo 2 Women will receive an oral placebo similar to dexketoprofen 2 hours before the procedure
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: dexketoprofen — Drug: dexketoprofen Women will receive oral dexketoprofen 25mg 2 hours before the procedure
  Drug: Placebo 1 Women will receive an oral placebo similar to Tramadol 2 hours before the procedure.
  Arms: dexketoprofen
Drug: Tramadol — Drug: Tramadol Women will receive oral Tramadol 100 mg 2 hours before the procedure
  Drug: Placebo 2 Women will receive an oral placebo similar to dexketoprofen 2 hours before the procedure
  Arms: tramadol
Drug: Placebo — Drug: Placebo 1 Women will receive an oral placebo similar to Tramadol 2 hours before the procedure.
  Drug: Placebo 2 Women will receive an oral placebo similar to dexketoprofen 2 hours before the procedure
  Arms: placebo

SUMMARY:
Two hundreds and twenty five postmenopausal women undergoing outpatient hysteroscopy and endometrial biopsy will be randomly divided into three equal groups. To ensure blinding the investigators will use the double dummy technique in which group 1 will receive Tramadol 100mg (Trama®, Global Napi, Giza, Egypt) orally in addition to a placebo similar to Celecoxib, group 2 will receive dexketoprofen 25mg (neo ketadex 25, Marcryl, Egypt) in addition to a placebo similar to Tramadol, and group 3 will received a placebo similar to Tramadol and a placebo similar to Celecoxib. All drugs will be given 2 hours before the procedure. An independent person will generate the allocation sequence using computer generated random numbers.

DETAILED DESCRIPTION:
Two hundreds and twenty five postmenopausal women undergoing outpatient hysteroscopy and endometrial biopsy will be randomly divided into three equal groups. To ensure blinding the investigators will use the double dummy technique in which group 1 will receive Tramadol 100mg (Trama®, Global Napi, Giza, Egypt) orally in addition to a placebo similar to Celecoxib, group 2 will receive dexketoprofen 25mg (neo ketadex 25, Marcryl, Egypt) in addition to a placebo similar to Tramadol, and group 3 will received a placebo similar to Tramadol and a placebo similar to Celecoxib. All drugs will be given 2 hours before the procedure. An independent person will generate the allocation sequence using computer generated random numbers.

Statistics:

Quantitative data will be statistically represented in terms of mean ± standard deviation (± SD) while categorical data will be represented as frequency and percentage. Comparison of quantitative data will be done using ANOVA test for independent samples while categorical data will be compared using Chi squared test or Fisher exact test when appropriate. A probability value (p value) less than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Post menopausal women.
* vaginal bleeding.
* Endometrial thickness >4mm.

Exclusion Criteria:

* Medical disorders like uncontrolled diabetes or hypertension, cardiac, renal, liver disease.
* Gastritis or peptic ulcer.
* Allergy to Tramadol or dexketoprofen.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Patient's perception of pain during the procedure | 2 minutes after starting the procedure
  The nurse will hand the patient a VAS and the patient will mark the point corresponding to her pain.VAS of 0 indicates no pain and VAS of 10 indicates the worst possible experienced pain

SECONDARY OUTCOMES:
Pain after the procedure | 30 minutes after completing the procedure
  The nurse will hand the patient a VAS and the patient will mark the point corresponding to her pain.

CONTACTS AND LOCATIONS:
Overall Officials: AHMED SAMY, MD, Principal Investigator — lecturer in obstetrics and gynecology,cairo university